CLINICAL TRIAL: NCT02581709
Title: The Development and Feasibility Testing of an Intervention Programme to Reduce Cognitive Impairment Due to Cancer Treatment
Brief Title: An Intervention Programme to Reduce Cognitive Impairment Due to Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very low recruitment and funding was unavailable to support further research.
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other); Cancer Research Network (Other)
Responsible Party: Principal Investigator, Michael Donnelly, Professor Michael Donnelly, Queen's University, Belfast
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STL/5086/14
Record Dates: First submitted 2015-10-15; First posted 2015-10-21 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Breast Neoplasms; Colorectal Neoplasms
Keywords: Feasibility study; Cognition; Chemotherapy; Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Countering cognitive impairment (Experimental): Each participant will complete neuropsychological assessments at baseline (prior to chemotherapy) and after chemotherapy. Patients identified as experiencing cognitive decline measured using Reliable Change Index on at least one cognitive function measure from before until after chemotherapy will be offered the intervention. Participants in the interventions will complete a neuropsychological assessment after completion of the intervention. Questionnaires to assess other non-cognitive factors e.g. quality-of-life will be administered at the end of chemotherapy to all participants and after the intervention to participants in the intervention.
  Interventions: Behavioral: Countering cognitive impairment

INTERVENTIONS:
Behavioral: Countering cognitive impairment — The intervention will include education about cancer-related cognitive impairment, instruction on relaxation techniques, compensatory techniques, goal-setting and lifestyle advice. Each session will last between 90 and 120 minutes, once a week for six weeks. The intervention will be delivered in a group setting, in a non-clinical environment by the investigators.

SUMMARY:
The goal of this research study is to test the feasibility of an intervention programme to reduce cognitive impairment due to cancer treatment. The investigators want to find out how acceptable the intervention and procedures are for cancer patients.

DETAILED DESCRIPTION:
The intervention programme will consist of the following components: education about cancer-related cognitive impairment, relaxation techniques, compensatory techniques, goal-setting and lifestyle advice. Each session will last between 90 and 120 minutes, once a week for six weeks. The intervention will be delivered in a group setting, in a non-clinical environment by the investigators.

The investigators aim to recruit 54 cancer patients from the local Cancer Centre onto the study. The cognitive functioning of cancer patients due to start chemotherapy will be assessed. Each patient's cognitive function will be reassessed after completion of chemotherapy and additional self-report measures will be administered. Patients who demonstrate cognitive decline over the course of chemotherapy will be invited to take part in the intervention programme. All other patients will be given an information sheet and advised to contact a member of their health-care team if they notice any changes in their cognitive function. The investigators aim to take 30 patients through the intervention. At the end of the intervention, each participant will complete an intervention evaluation questionnaire in addition to the cognitive functioning assessments and self-report measures.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* Have a diagnosis of early stage breast or colorectal cancer (Stage I-III disease)
* Are planned to receive standard care adjuvant chemotherapy.
* Able to complete Neuropsychological test assessment pre- and post- chemotherapy receipt.
* Proficiency in the English language
* Able to provide informed consent
* Patients with breast cancer can be receiving standard care hormonal therapy or radiotherapy

Exclusion Criteria:

* Treatment plan does not include chemotherapy.
* Diagnosed with metastatic cancer
* Treatment plan includes cranial radiation, brain surgery or intrathecal therapy.
* History of previous cancer, as previous treatment or experience may contribute to cognitive impairments (with the exception of non-melanoma skin cancer).
* History of cranial radiation, brain surgery or intrathecal therapy due to the direct impact on the brain.
* History of, or, comorbid condition which may alter cognitive function tests i.e. stroke, head injury, epilepsy, Parkinson's disease, Huntington's disease, Alzheimer's disease, encephalitis, substance abuse, bipolar disorder, psychosis, schizophrenia and learning disability.
* Current use of psycho-stimulant medication e.g. Methylphenidate which increases activity in the central nervous system, or central nervous system (CNS) depressant medication e.g. Benzodiazepines and Barbiturates due to slowing down of cognitive processes. Use of commonly prescribed anti-depressants e.g. Monoamine Oxidase Inhibitors (MAOIs), Selective Serotonin Reuptake Inhibitors (SSRIs) or Serotonin Noradrenaline Reuptake Inhibitors (SNRIs) or Tricyclic Antidepressants (TCAs) is permitted.
* Have a Mini-Mental Status Examination score ≤23 indicative of substantial cognitive impairment including dementia.
* Current uncontrolled mood disorder e.g. Major depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention implementation | After 27 weeks
  The investigators aim to assess the acceptability of the intervention programme and its procedures to patients enrolled in the study. This is a non-validated questionnaire designed specifically for this study. Participants are required to rate the verbal and written information about the study, advice about the study, overall intervention, specific intervention components, each assessment visit and procedure, length of time of intervention and assessment visits on a three- or five-point likert scale. Open-ended questions asking participants to provide further information were provided.

SECONDARY OUTCOMES:
Hopkins Verbal Learning Test | At baseline, after chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to capture memory and learning. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Reitan's Trail Making Test (TMT) A and B | At baseline, after chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to capture executive functions and visuomotor speed. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Controlled oral Word Association (COWA) sub-test of the Multilingual Aphasia Examination | At baseline, after chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to capture executive functions and verbal ability. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Neuropsychological Assessment Battery Digit Span sub-test | At baseline, after chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to capture working memory and attention. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
STROOP test | At baseline, after chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to capture attention. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Functional Assessment of Cancer Therapy- Cognitive Subscale (FACT-Cog) | After chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to self-reported cognitive function. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Short form health survey (SF-36) | After chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to self-reported health-related quality of life. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Centre for Epidemiological studies Depression- Revised scale (CESD-R) | After chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to self-reported depression. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Hospital Anxiety and Depression Scale- Anxiety sub-scale (HADS-A) | After chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to measure state anxiety. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Functional Assessment of Chronic Illness Therapy- Fatigue sub-scale (FACIT-F) | After chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to measure self-reported fatigue. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Pittsburgh Sleep Quality Index (PSQI) | After chemotherapy (15 weeks since baseline assessment for breast cancer patients and 21 weeks since baseline for colorectal cancer patients) and after the intervention (approximately 27 weeks from baseline assessment).
  This test is used to measure self-reported sleep disturbances. As this is a feasibility study this measure is not used to assess the effectiveness of the intervention and only means and standard deviations will be calculated.
Cognitive Reserve Scale | Before Chemotherapy
  This scale is used to capture engagement in cognitive activities throughout the lifespan.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnelly, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Cancer Centre, City Hospital, Belfast HSC Trust, Belfast, Antrim, United Kingdom